CLINICAL TRIAL: NCT07292701
Title: Impact of Kinesiotaping Application on Pelvic Girdle Pain in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Walaa Ibrahim mohamed abdou, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005903
Record Dates: First submitted 2025-12-06; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Pelvic Girdle Pain; Kinesiotaping; Pregnancy Complications
MeSH Terms: conditions — Pelvic Girdle Pain; Pregnancy Complications | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- core exercise (Experimental): It included 24 women who will be treated by doing core exercise only.
  Interventions: Other: Core stability exercises
- kinesiotaping (Active Comparator): It will include 24 women who will be treated by applying kinesiotaping for 5 days twice in two consecutive weeks with core exercise
  Interventions: Other: Kinesio tape
- adhesive tape (Active Comparator): It will include 24 women who will be treated by applying adhesive tape instead of kinesiotape for 5 days twice in two consecutive weeks with core exercise.
  Interventions: Other: Kinesio tape; Other: Core stability exercises

INTERVENTIONS:
Other: Kinesio tape — Kinesio taping is a drug-free elastic therapeutic technique developed by Dr. Kenso Kase in the 1970s, utilized for treating various musculoskeletal issues, including pain and dysfunction. It is known for having no side effects, contributing to its popularity among practitioners. In a study, participants underwent five days of Kinesio taping applied by the same therapist, focusing on the lumbar region of pregnant women. The tape used was an elastic, waterproof material that allows for motion, applied in specific vertical and horizontal configurations to alleviate lumbar and pelvic girdle pain.
  Arms: adhesive tape; kinesiotaping
Other: Core stability exercises — All participants will do core exercise. The control group (Group A) received no additional treatment. The core exercises were in form exercises that promote bracing or excessively increasing trunk muscle activation Popular core stability exercise programs commonly focus on bracing or activating the trunk muscles that are believed to support the spine. This includes exercises such as: crunches, planks, bird-dogs
  Arms: adhesive tape; core exercise

SUMMARY:
The aim of this study is to determine the effect kiensio taping in relieving pelvic girdle pain during pregnancy in terms of decrease pain and improving function and quality of life.

DETAILED DESCRIPTION:
Severity of pelvic girdle pain can be different, as a result of the progress of the disorders and subjective feeling of pain. According to Kanakaris an average severity of pain in pelvic girdle pain is 50-60 mm scale visual analogue scale. Results may vary according to different factors such as; pregnancy stage, age of the pregnant women, different body mass index. Beyond the discomfort and pain, pelvic girdle pain can also limit the performance of the activities of daily living such as; bending, lifting, sitting, sleeping, housework, long walking, and standing and thus adversely affect the quality of life of pregnant women. Unfortunately, the options for pain therapy in pregnant women are significantly limited due to the possible danger to both mother and fetus. Most of the standard drugs used affect the fetus and are not recommended, especially for long-term treatment.

There is very little clinical experience and only limited documentation for effectiveness of Kinesio taping on pelvic girdle pain during pregnancy. Because the existing treatments for pregnancy-related pelvic girdle pain are not adequately known and are not found to be reliable by patients and clinicians. Kinesio taping may be a potential treatment if it is an effective and tolerable method. Therefore, the aim of the present study was to determine the influence of Kinesio taping pelvic girdle pain in pregnant women

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-36 years old.
* Gestational age: 10-34 week of pregnancy.
* Low back pain experienced anywhere from T12 to the gluteal fold without leg pain, and at least moderate pain intensity (scoring ≥4 on visual analogue scale)
* At least one positive test out of three applied, which are Long Dorsal Ligament Test (modified for pregnant women), Posterior Pelvic Pain Provocation (4P), and Trendelenburg test (modified for pregnant women).
* Negative Straight Leg Raise test

Exclusion Criteria:

* History of abortion
* pregnancy of twins
* previous of pelvic injury.
* Skin previous injury in the lumbosacral area.
* Positive Straight Leg Raise test
* Negative diagnostic tests for pelvic girdle pain
* Chronic pelvic diseases.
* History of allergies to material of kinesiotape.

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
assessment of pain intensity | At baseline and after 2 weeks
  Visual Analogue Scale (VAS) is a widely used method for assessing pain intensity, functioning as a subjective measure of treatment efficacy. It involves marking a point on a 10-cm line that indicates pain levels from "no pain" to "worst pain." Studies validate VAS as a reliable interval scale for measuring both acute and chronic pain, making it a useful tool in clinical practice. Pain levels are measured before and after 5 days of treatment, followed by another recording after re-application of the tape after an additional 5 days.

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, faculty of physical therapy, Cairo university, Cairo, Egypt